CLINICAL TRIAL: NCT05288374
Title: Celecoxib for Treatment of Postoperative Pain After Osteosynthesis of Distal Radius Fracture
Brief Title: Celecoxib in Postoperative Analgesia for Radius Fracture Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Jiri Malek, Assoc. Prof. Jiri Malek, MD, Ph.D., Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Celecoxib in radius fracture
Record Dates: First submitted 2022-03-10; First posted 2022-03-21 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Pain, Postoperative
Keywords: Postoperative pain; Distal radius fracture; Osteosynthesis; Celecoxib
MeSH Terms: conditions — Pain, Postoperative; Wrist Fractures | interventions — Celecoxib

STUDY DESIGN:
Intervention Model Description: Celecoxib 100 mg orally on the day of surgery at 6 in the morning and will be continued regularly at 6 in the morning and 6 in the afternoon for 3 days.
Who Masked: Participant
Masking Description: Placebo pill provided by a hospital pharmacy will be administered orally on the day of surgery at 6 in the morning and will be continued regularly at 6 in the morning and 6 in the afternoon for 3 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Celecoxib (Experimental): Celecoxib 100 mg orally will be administered in the day of surgery at 6 in the morning and will be continued regularly at 6 in the morning and 6 in the afternoon for 3 days.
  Interventions: Drug: Celecoxib 100 mg
- Placebo (Placebo Comparator): A placebo pill provided by a hospital pharmacy will be administered in the day of surgery at 6 in the morning and 6 in the afternoon for 3 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib 100 mg — Administering Celecoxib 100 mg (Celebrex) regularly every 12 hours for 3 days starting at 6 in the morning on the day of surgery
  Other Names: Celebrex 100 mg
  Arms: Celecoxib
Drug: Placebo — Administering placebo regularly every 12 hours for 3 days starting at 6 in the morning on the day of surgery
  Other Names: Placebo pill
  Arms: Placebo

SUMMARY:
Patients scheduled for elective osteosynthesis of the distal radius will be randomized to receive celecoxib 100 mg orally (PO) at 6 in the morning before surgery and every 12 hours for 2 days thereafter, or a placebo pill in the same regimen. After surgery under general anaesthesia, they will receive paracetamol 1 g intravenously (IV) every 6 hours and if pain intensity is greater than 4 on a numeric rating scale (NRS) of 0-10, piritramid 15 mg intramuscularly (IM) will be administered. Pain intensity, piritramid consumption and side effects of treatment will be recorded in a questionnaire for 2 days.

DETAILED DESCRIPTION:
A prospective single-blinded randomized study will be performed in patients of the Orthopaedic Clinic of the 3rd Medical Faculty of Charles University (3LF UK) and the Faculty Hospital Kralovske Vinohrady (FHKV) scheduled for elective osteosynthesis of the distal radius. The expected number of participants is 25 in each arm of the study. They will be randomized by envelope method into an non-steroidal analgesic (NSA) group, which will receive celecoxib at 6 in the morning before surgery, and a C group, which will receive a placebo pill prepared by the hospital pharmacy. General anesthesia will be performed in both groups in the standard way using propofol, sufentanil and sevoflurane 1 minimal alveolar concentration (MAC) with air and oxygen at 40% concentration. At the end of surgery, each patient will be given paracetamol 1 g intravenously (IV) and ondansetron 4 mg IV. Pain intensity after surgery will be measured on a numerical rating scale (NRS) 0-10. For postoperative analgesia, both groups will receive paracetamol 1 g IV. every 6 hours, and for NRS>4 pain intensity, piritramid 15 mg intramuscularly (IM). The NSA group will receive celecoxib 100 mg orally (PO) at 6 in the morning and 6 in the afternoon, and group C will receive placebo at the same interval.

Parameters to be monitored will be postoperative pain intensity for the primary objective, and opioid piritramid consumption and side effects of the treatment for the secondary objectives. NRS, number of doses of piritramid and side effects will be recorded in a coded questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for osteosynthesis of distal radius fracture

Exclusion Criteria:

* Known hypersensitivity (e.g., anaphylactic reactions and serious skin reactions) to celecoxib
* History of asthma, urticaria, or other allergic-type reactions after taking aspirin or other NSAIDs.
* Patients who have demonstrated allergic-type reactions to sulfonamides.
* Inability to understand the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity | up to 2 days
  Intensity of pain measured by numeric rating scale (NRS) 0-10

SECONDARY OUTCOMES:
Number of piritramid injection | 3 days
  Piritramid 15 mg intramuscularly will be administered if numeric rating scale (NRS 0-10) of pain is NRS>4
Side effects of treatment | 3 days
  Incidence of stomach pain, heartburn, gas, diarrhea, constipation, nausea, vomiting, dizziness, others

CONTACTS AND LOCATIONS:
Overall Officials: Jiří Málek, MD, Principal Investigator — 3rd Medical Faculty of Charles University and Faculty Hospital Kralovske Vinohrady
Locations (2):
- Czechia (2):
  - Faculty Hospital Kralovske Vinohrady, Prague
  - Jiří Málek, Prague